CLINICAL TRIAL: NCT02689167
Title: Open Label, Randomised Multi-centre Phase II Study to Assess the Efficacy and Tolerability of Sunitinib by Dose Administration Regimen (Dose Modification or Dose Interruptions) in Patients With Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Study to Assess Various Sunitinib Schedules in Renal Cell Carcinoma
Acronym: SURF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2015/254
Record Dates: First submitted 2016-02-10; First posted 2016-02-23 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Kidney Neoplasms; Metastatic Renal Cell Cancer
Keywords: renal cell carcinoma; sunitinib; metastatic; schedule; toxicity; safety
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A 4/6 (Active Comparator): Sunitinib 37.5 mg/day; regimen 4/6 (Marketing Authorisation Indication) 4 weeks "on " alternating with 2 weeks "off "
  Interventions: Drug: Sunitinib
- Arm B 2/3 (Experimental): Sunitinib 50 mg/day; regimen 2/3 (experimental arm) 2 weeks "on " alternating with 1 week "off "
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib

SUMMARY:
Patients who are candidates for first line treatment with Sunitinib 50mg 4/6 regimen in accordance with the Marketing Authorisation who meet the inclusion/exclusion criteria will be offered participation in this study during the consultation as part of their usual care. The patients will be included before Sunitinib treatment is started. Thereafter, sunitinib is initiated 50 mg/day; regimen 4/6 (Marketing Authorisation Indication), 4 weeks "on " alternating with 2 weeks "off "

As soon as a dose or schedule adjustment is required, regardless of cause, the patient will be randomised 1/1:

* Either into arm A and will receive 37.5mg of Sunitinib per day by the 4/6 regimen (in accordance with the Marketing Authorisation); 4 weeks "on " alternating with 2 weeks "off "
* Or into arm B and will receive 50mg of Sunitinib per day by the 2/3 regimen (investigational arm); 2 weeks "on " alternating with 1 week "off "

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women over 18 years old
* Patients with local, advanced or inoperable or metastatic (MRCC) renal cell carcinoma who are starting first line treatment with Sunitinib 50mg (4/6 regimen) according to the Marketing Authorisation Indication
* Patients with histologically or cytologically confirmed renal cancer, clear cell variant or with a clear cell component
* Karnofsky performance status ≥ 70%
* Adequate organ function:

  * Absolute neutrophil (N) count ≥ 1 500 / µL
  * Platelets ≥ 100 000 / µL
  * Haemoglobin ≥ 10 g/dL
  * Adjusted serum calcium ≤ 2.6 mmol/L
  * Creatinine clearance ≥ 30 mL/min (by the MDRD formula)
  * Total bilirubin ≤ 1.5 x ULN (upper limit of the normal range)
  * AST ≤ 2.5 x ULN and ALT ≤ 2.5 x ULN OR AST and ALT ≤ 5 x ULN if liver abnormalities due to liver metastases AST = aspartate aminotransferase ALT = alanine aminotransferase

Key Exclusion Criteria:

* Renal carcinoma with no clear cell component.
* Previous systemic treatment for the RCC regardless of type (including targeted therapy, immunotherapy, chemotherapy, hormone or experimental therapy). Previous or concomitant treatment with a bisphosphonate or denosumab is allowed.
* Patients whose clinical state and comorbidities are not consistent with administration of Sunitinib at the initial dose of 50mg/day 4 weeks out of 6.
* Grade 3 haemorrhage within 4 weeks before starting treatment with Sunitinib (according to the NCI-CTCAE toxicity score version 3.0).
* The presence of a past history of cancer in the 3 years before inclusion into the study
* Major surgery within 4 weeks before sunitinib initiation
* Past history of symptomatic cerebral metastases, spinal cord compression or meningeal carcinomatosis. Patients with cerebral metastases discovered incidentally on imaging and who are asymptomatic are not excluded if these metastases have been treated (radiotherapy and/or surgery) with a period of at least 4 weeks between the end of treatment and inclusion into the study and no clinical or radiological signs of relapse, and corticosteroid dose is not exceeding 10mg/day of prednisone or equivalent. Subjects will be excluded if subjects have signs of grade ≥ 2 treatment-related complications.
* Any of the following features within 6 months of the administration of Sunitinib: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
* Pulmonary embolism or deep vein thrombosis within 3 months of inclusion (unless it's stable, asymptomatic and treated with a low molecular weight heparin for at least 6 weeks before inclusion).
* Any known acute or chronic disorder (such as severe chronic obstructive pulmonary disease) which in the opinion of the investigator could impact on the patient's capacity to receive the study treatment or make interpretation of toxicity or adverse events difficult.
* Known HIV infection.
* History of chronic active hepatitis including subjects who are carriers of the hepatitis B (HBV) or hepatitis C (HCV) virus.
* Existence of uncontrolled infection.
* Uncontrolled hypertension defined as a blood pressure of > 150 mmHg systolic or > 100 mmHg diastolic despite optimal anti-hypertensive therapy (blood pressure must be controlled at inclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
MDT (median duration of treatment) | 12 mo
  The primary objective of this study is to estimate the median duration of treatment in each treatment group (arm A vs arm B) calculated from sunitinib initiation.

SECONDARY OUTCOMES:
PFS (progression-free survival) | 12 months
  To estimate progression-free survival in patients included in each of the groups and in the overall population included in this study.
OS (overall survival) | 30 months
  To estimate overall survival in patients included in each of the groups and in the overall population included in this study.
duration of sunitinib post randomization | 12 months
  Estimation of the time between date of randomization and sunitinib arrest (for any reason) in the two treatment arms.
time to randomization | 4 months
  To estimate the time to randomization defined as the time between the date of sunitinib initiation and the date of randomization.
ORR (objective response rate) | 6 months
  To measure the objective response rate according to RECIST 1.1 criteria.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
  To assess safety profile before and after randomization.
QOL (quality of life) | 24 months
  To assess health-related quality of life since sunitinib is started (before randomization, at the time of randomization and after randomization)

CONTACTS AND LOCATIONS:
Overall Officials: antoine thiery-vuillemin, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mouillet G, Paillard MJ, Maurina T, Vernerey D, Nguyen Tan Hon T, Almotlak H, Stein U, Calcagno F, Berthod D, Robert E, Meurisse A, Thiery-Vuillemin A. Open-label, randomized multicentre phase II study to assess the efficacy and tolerability of sunitinib by dose administration regimen (dose modification or dose interruptions) in patients with advanced or metastatic renal cell carcinoma: study protocol of the SURF trial. Trials. 2018 Apr 12;19(1):221. doi: 10.1186/s13063-018-2613-8. PMID 29650037